CLINICAL TRIAL: NCT04924920
Title: Sigh35 and End-expiratory Occlusion Test (EEOT) for Assessing flUid Responsiveness in Critically Ill Patients Undergoing Pressure Support Ventilation
Acronym: SETUP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Humanitas Clinical and Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SIGH_EEOT
Record Dates: First submitted 2021-06-04; First posted 2021-06-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Critically Ill Patients; Hemodynamic Instability; Mechanical Ventilation Pressure High

STUDY DESIGN:
Intervention Model Description: Cross-over design. The study has one single arm cross-over treatment design. The same patient will be assessed by means of the two tests. The sequence of application will be randomly generated and applied to the patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention EEO_SIGH (Experimental): Single arm intervention. All the patients will receive the two tests (SIGH and EEOT) in 1:1 random sequence order
  Interventions: Diagnostic Test: SIGH; Diagnostic Test: EEOT; Diagnostic Test: Fluid challenge

INTERVENTIONS:
Diagnostic Test: SIGH — To add the Sigh35 to PSV, the ventilator is set in pressure controlled synchronized intermittent mandatory ventilation plus PSV [SIMV (PC) + PS mode], with SIMV rate set a 1/min and inspiratory time of 4 seconds. SIMV (PC) = 35 cmH20 of total inspiratory support (PEEP + PS).
Diagnostic Test: EEOT — • The EEOT is performed by interrupting the mechanical ventilation for 15 seconds, by using and end-expiratory hold on the ventilator. The ventilator trigger is set at 2 L/min.
Diagnostic Test: Fluid challenge — Bolus of fluids of 4 ml/kg given within 10 minutes

SUMMARY:
The application of a brief SIGH of 4 seconds at 35 cmH20 has shown to reliably predict fluid responsiveness in critically ill patients undergoing pressure support ventilation.

The end-expiratory occlusion test (EEOT) has been also used in the same type of patients, with the same purpose, but in a limited amount of studies.

The aim of this study is to compare the reliability of the the two test in assessing fluid responsiveness.

DETAILED DESCRIPTION:
Assessing preload dependence in critically ill patients is a challenge for the Intensive Care Unit (ICU) physicians. During controlled mechanical ventilation, dynamic indexes can be applied in non-arrhythmic patients with sufficiently high tidal volume (VT), i.e., >8 ml/kg and non-severely impaired lung compliance. The interplay between mechanical ventilation and hemodynamic is more complex in patients with a spontaneous breathing activity, whose respiratory efforts affect intrathoracic pressure and venous return to the right ventricle (RV).

To overcome these limitations, functional hemodynamic assessment, consisting in maneuvers determining a sudden change in cardiac preload, such as Passive leg raising (PLR) or end-expiratory occlusion test (EEO), represents a valuable means for assessment of fluid responsiveness.

Both PLR and EEO have been successfully utilized for assessing fluid responsiveness, regardless of ventilatory assistance and mode of ventilation. Unfortunately, however, some drawbacks limit the extensive use of these maneuvers in clinical practice. One the one hand, PLR cannot be applied in some clinical situations, such as traumatisms of the hip, legs or lumbar spine, deep venous thrombosis, intracranial or abdominal hypertension. Indeed, a recent large observational study showed PLR to be the most common form of assessment of fluid responsiveness, being used, nonetheless, in only 10.7% of the patients necessitating the assessment of fluid responsiveness. On the other hand, rates of EEO failure as high as 22.5 % have been reported, consequent to visible patient's effort against the occluded airway.

It has been recently successfully tested a new approach for assessing fluid responsiveness in patients undergoing partial ventilatory assistance. It has been proposed that the changes from baseline of systolic arterial pressure (SAP), pulse pressure (PP) and stroke volume index (SVI) in relationship to the airway pressure (Paw) generated during a "sigh" maneuver can predict fluid responsiveness in ICU patients undergoing pressure support ventilation (PSV) In the first "proof of concept" study (performed in 40 hemodynamically unstable ICU patients) three sighs has been tested, in a computer-generated random order, at either 15 (SIGH15), 25 (SIGH25) and 35 (SIGH35) cmH2O of total inspiratory Paw (PEEP + PSV). The results showed that only the variation of the pulse pressure recorded after SIGH35 application successfully predicted fluid responsiveness. [AUC of PP after SIGH35 = 0.91 (0.82 - 0.99); sensitivity 75% (47.6%-92.7%) and specificity 91.6 (73.0%- 98.9%); best threshold value of the ROC curve was -35% from baseline].

Hemodynamic Measurements. All patients will be equipped with a continuous hemodynamic monitoring of arterial waveform.

The primary end point will be assessed by means comparison of the areas (AUC) under receiver operating characteristic (ROC) curves: considering the data reported in the literature, we assumed that the AUC of the SIGH35 should be of at least 0.85 to be clinically relevant. This value was compared to the null hypothesis (AUC = 0.65; ratio of samples sizes in negative and positive groups of 1:1): the calculated sample size is 50 patients. Considering the possibility of the occurrence extrasystoles during the beat-to-beat evaluation of the EEOT and the SIGH, the sample size is inflated by the 20% to account for the rate of loss of patients during the post-hoc data analysis. The final sample size is 60 patients.

Fluid responsiveness is defined as a CI increase ≥ 10% after FC infusion.

ELIGIBILITY:
* Adult (>18 yo) ICU patients undergoing PSV ventilation
* Inspiratory support level (PS) between 8 and 15 cmH2O and positive end-expiratory pressure (PEEP) between 5 and 12 cmH2O,
* Presence of acute circulatory failure defined as:

  * Systolic blood pressure (SBP) ≤90 mmHg or mean arterial pressure (MAP) ≤70 mmHg or requiring vasopressors to maintain SBP >90 mmHg or MAP >70 mmHg or decline of SBP > 50 mm Hg in known hypertensive patients, along with one or more of the following:
  * urinary flow ≤0.5 mL/kg/min for ≥2 hours
  * heart rate ≥100 beats per minute
  * presence of skin mottling and 4) blood lactate concentration ≥4 mmol/L.

Exclusion criteria

* left ventricular ejection fraction <30% or severe valvular dysfunction
* atrial fibrillation
* severe acute respiratory distress syndrome (ARDS)
* abdominal compartment syndrome
* air leakage through chest drains
* artifacts in arterial waveform
* pathological respiratory patterns due to neurological diseases
* signs of fatigue or respiratory distress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Pulse pressure prediction of fluid responsiveness | Evaluated before and after SIGH35 (within 1 minute from SIGH35 application)
  Pulse pressure changes after SIGH35 application
Stroke volume prediction of fluid responsiveness | Evaluated before and after SIGH35 (within 1 minute from SIGH35 application)
  Stroke Volume changes after SIGH35 application

SECONDARY OUTCOMES:
Pulse pressure prediction of fluid responsiveness | Evaluated before and after EEOT (within 1 minute from EEOT application)
  Pulse pressure changes after EEOT application
Stroke volume prediction of fluid responsiveness | Evaluated before and after EEOT (within 1 minute from EEOT application)
  Stroke Volume changes after EEOT application

OTHER OUTCOMES:
Rate of failure of SIGH test | During the test execution
  Presence of cough
Rate of failure of EEOT test | During the test execution
  Trigger of the ventilator

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analyzed during this study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Messina A, Colombo D, Barra FL, Cammarota G, De Mattei G, Longhini F, Romagnoli S, DellaCorte F, De Backer D, Cecconi M, Navalesi P. Sigh maneuver to enhance assessment of fluid responsiveness during pressure support ventilation. Crit Care. 2019 Jan 28;23(1):31. doi: 10.1186/s13054-018-2294-4. PMID 30691523
- [Background] Patroniti N, Foti G, Cortinovis B, Maggioni E, Bigatello LM, Cereda M, Pesenti A. Sigh improves gas exchange and lung volume in patients with acute respiratory distress syndrome undergoing pressure support ventilation. Anesthesiology. 2002 Apr;96(4):788-94. doi: 10.1097/00000542-200204000-00004. PMID 11964584
- [Background] Monnet X, Osman D, Ridel C, Lamia B, Richard C, Teboul JL. Predicting volume responsiveness by using the end-expiratory occlusion in mechanically ventilated intensive care unit patients. Crit Care Med. 2009 Mar;37(3):951-6. doi: 10.1097/CCM.0b013e3181968fe1. PMID 19237902